CLINICAL TRIAL: NCT05536167
Title: Prospective Multicenter Study to Characterize the REAL-WORLD EVIDENCE Regarding Safety and Performance of the Aspiration Catheters Family
Status: Completed | Type: Observational
Sponsor: Arthesys (Industry)
Responsible Party: Sponsor
Other Study IDs: ART-ASPI CATHETER-01
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Thrombus in the Central and Peripheral Circulatory System, Including Saphenous Vein Grafts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this post market study is to collect clinical data of the Arthesys Aspiration catheters family during percutaneous intervention and/or stenting procedure of vessels in the central and peripheral circulation system, including saphenous vein grafts, to support MDR submission.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included as per Instructions for Use (IFU), Hospital standard of care and Good Clinical Practice (GCP):

  1. Patient with a percutaneous intervention to a native coronary, saphenous vein graft, or peripheral arteries;
  2. Patient with angiographic evidence of thrombus;
  3. Patient > or = 50 kg;
  4. Patient >18 years;
  5. Patient who understands the trial requirements and the treatment procedures and provides written informed consent.

Exclusion Criteria:

* Patients will be excluded as per IFU, Hospital standard of care and GCP, also if there are under judicial protection, guardianship or curatorship or if they are deprived of their liberty by judicial or administrative decision.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing PTA/PTCA and/or stenting procedures and presenting thrombus in the central and peripheral circulatory system, including saphenous vein grafts.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint | up to end of procedure
  successful debris aspiration (macroscopic observation of the retrieved material in the filter) during the procedure.
Safety endpoint | up to end of procedure
  insertion and retrieval of the catheter up to the treated vessel without complication.

SECONDARY OUTCOMES:
Performance - TIMI flow grade | up to end of procedure
  Final Thrombolysis In Myocardial Infarction (TIMI) Flow Grade at procedure
Safety - absence of complications | up to end of procedure
  Absence of complications during hospitalization (per standard hospital of care): cardiovascular death, recurrent myocardial infarction, cardiogenic shock, worsening of TIMI flow due to aspiration catheter, new or worsening New York Heart Association (NYHA) Class IV heart failure,
Performance - TIMI thrombus grade | up to end of procedure
  Final TIMI Thrombus Grade at procedure
Performance | up to end of procedure
  Distal Embolization Rate at procedure
Safety - absence of Serious Adverse Event | up to end of procedure
  Incident of Device Related SAEs during aspiration catheter use
Safety - absence of stroke | up to end of procedure
  Stroke during aspiration catheter use (per hospital standard of care).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Louis, La Rochelle, France